CLINICAL TRIAL: NCT06872736
Title: Innovative Use of Wereable Technology for Improving Functionality in Children with Unilateral Cerebral Palsy
Brief Title: Wereables for Upper Limb Functionality in Hemiparesis
Acronym: WeFun
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universidade da Coruña (Other)
Collaborators: Complexo Hospitalario Universitario de A Coruña (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PID2021-126782OA-I00; PID2021-126782OA-I00 (Other Grant/Funding Number: MCIN/AEI/ 10.13039/501100011033, by "ERDF A way of making Europe")
Record Dates: First submitted 2025-02-10; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2024-03

CONDITIONS: Unilateral Cerebral Palsy
Keywords: children; unilateral cerebral palsy; function; mobility; upper limb; weareable; technology; routines; family centered approach; activity; participation; family; developmental disregard; environmental enrichment; natural environment; quality of life; movement analysis; fatigue; upper extremity; family involvement in research; hemiparesis; cerebral palsy; early intervention
MeSH Terms: conditions — Motor Activity; Fatigue; Paresis; Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Selected Physical Therapy Program, wearable, routine program, double blind, contrabalanced randomization
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Allocation in the experimental and control group is blinded for children, families and researchers who assesses. Outcome measures are blinded for the researcher doing the intervention. Researchers doing the analysis are blinded to the conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1 month daily routine program with wefun-weareable activated (Experimental): Children will follow a daily routine program based on goals set by families, which will be initiated by the wearable. Children in the experimental group will have the wearable's experimental movement functions activated.
  Interventions: Device: WeFun-wearable activated
- 1 month daily routine program with wefun-wearable desactivated (Active Comparator): Children will follow a daily routine program based on goals set by families, which will be initiated by the wearable. Children in the control group will not have experimental functions in their wearables.
  Interventions: Device: WeFun-wearable desactivated

INTERVENTIONS:
Device: WeFun-wearable activated — 1 month daily routine program with weekly visits in natural environments (home, community, etc) together with WeFun-weareable to increase spontaneous use of the upper limb in children with UCP during activities of daily life and leisure. Activities are priorized by Canadian Occupational Performance Measure and Goal Atteinment Scale. Programs are designed together with a transdisciplinary team, acting as consultants. Children in the experimental group will have the wearable's experimental movement functions activated.
  Arms: 1 month daily routine program with wefun-weareable activated
Device: WeFun-wearable desactivated — 1 month daily routine program with weekly visits in natural environments (home, community, etc) together with WeFun-weareable to increase spontaneous use of the upper limb in children with UCP during activities of daily life and leisure. Activities are priorized by Canadian Occupational Performance Measure and Goal Atteinment Scale. Programs are designed together with a transdisciplinary team, acting as consultants. Children in the control group will not have experimental functions in their wearables.
  Arms: 1 month daily routine program with wefun-wearable desactivated

SUMMARY:
The project is configured as a national interventional study that aims to determine the effectiveness of an intervention strategy using wearable technology, tailored to improve function (WeFun-wearable), on the spontaneous use of the affected upper extremity, activities of daily living and the participation in children with unilateral cerebral palsy.

DETAILED DESCRIPTION:
Cerebral palsy represents the most common paediatric neurological disorders. Unilateral cerebral palsy (UCP) subtype is the most frequent, accounting for about 0.6-1 per 1000 live births. Many children with UCP experience upper limb dysfunction, which is often more pronounced than that on lower extremity limitation. Rehabilitation strategies on the affected upper limb are of paramount importance to diminish limitations, especially those that seek to improve independence and wellbeing. These strategies are often provided through technology, which got into the clinics spotlight years ago, after extensive innovation-driven and knowledge research.

However, technology development has not reached its tops and technology solutions will drive the optimization of scientific evidence-based rehabilitation strategies. In this project, we use scientific knowledge acquired in our laboratory regarding the validation of new technologies to evaluate and treat movement disorders. Specifically, an unprecedented wearable will be used that could assess movement and complement intervention to influence function to such an extent that it would ultimately improve participation and quality of life for children with UCP.

WeFun proposes a home-based multimodal technology-based training, related to the practice of activities of daily life, to improve the use of the affected upper limb. WeFun wearable allows daily assessment of the amount of movement, in combination with training of upper limb movements and daily routines for children with CP. Our hypothesis is that a wearable technology to improve function, the We-Fun-wearable, could be an effective tool for the assessment and approach of the upper limb in children with CP.

This study has the potential to establish a new evidence-based and cost-effective therapy, accessible to children with cerebral palsy and their families, so that a digital solution can be provided for a vulnerable group: children with disabilities.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of UCP.
* Children aged between 3 and 8 years old.
* Children rated on levels I to III on the Manual Ability Classification System (MACS).

Exclusion Criteria:

* Botulinum toxin injection or surgical interventions in the upper limb within 6 months prior to study entry.
* Medical complications non-controlled that would interfere with study participation (e.g., not controlled epilepsy).
* Predominantly athetoid or dystonia movement patterns.
* Insufficient cognitive level to follow instructions,
* Non-corrected marked visual impairments.

Families can be retired from the study after starting if:

* Families don't assist or don't collaborate in the weekly sessions with the reference person.
* Wearable activity if presumably lower than expected (few recordings of activity, <20%).
* Families don't provide feedback about daily sessions through the satisfaction system in the app/registration sheet.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-06-07 (Actual); Primary Completion 2024-09-14 (Actual); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Bimanual performance/functional hand use | Baseline, immediately after the intervention and after 2 months follow-up
  The Assisting Hand Assessment (AHA) evaluates the spontaneous use of the more affected upper limb during bimanual activities. For these assessments a semi-structured play session with standardized toys and materials, that require the use of both hands, is performed and video-recorded. Subsequently, 20 items are scored in a rating range of 4 points, and the sum of scores in AHA may vary between 22 and 88 points. Through Rasch analysis this ordinal scale is transformed into AHA units ranging from 0 to 100 to obtain the final score. The AHA has shown to be a reliable and valid assessment for children and adolescents with unilateral cerebral palsy.

SECONDARY OUTCOMES:
Sociodemographic variables | Baseline, immediately after the intervention and after 2 months follow-up
  Those sociodemographic and clinical variables that may influence the data obtained will be recorded. These are: age, sex, medical diagnosis, therapeutic and medical interventions performed, manual ability classification system (MACS) level, medical complications, medication and vision/hearing/behavioral problems.
Upper Extremity Use (UEU) - WeFUN-wearable measure | Baseline, during intervention period, immediately after the intervention and after 2 months follow-up
  Activity recorded across six axes of the accelerometer and gyroscope of the wearable will be combined and processed to obtained Upper Extremity Use (UEU) variable which will represent the quantity of upper extremity movement (mean activity counts per second over an entire monitored activity). This activity will be recorder during all the protocol (assessments and intervention period).
Asymmetry Index (AI) - WeFUN-wearable measure | Baseline, immediately after the intervention and after 2 months follow-up
  During AHA assessment, UEU will be extracted separately for both the dominant and non-dominant (or affected) hand and calculated an Asymmetry Index (AI) following the Edinburgh Inventory formula to check how much each arm contributes to the activity. This measurement will be recorded only at the laboratory assessments.
Grip strength | Baseline, immediately after the intervention and after 2 months follow-up
  Grip strength is assessed with Biometrics E-LINK H-500 Hand Kit (dynamometer).
  children performed three MVC with the grip dynamometer with each hand. After each MVC, a 30-s rest was provided. The mean of the three trials is used.
Static motor fatigability | Baseline, immediately after the intervention and after 2 months follow-up
  Assessed with Biometrics E-LINK H-500 Hand Kit (dynamometer).
  Static motor fatigability will be measured during a 30-second sustained maximal contraction using the grip dynamometer. This measurement will be repeated three times.
  Static motor fatigability will be quantified with 2 outcome measures: mean force (Fmean) and the static fatigue index. First, the peak force within the first 10 seconds was identified, and only the curve after this peak was used in the calculations.
  For Fmean, the remaining time was divided into 3 equal parts, and Fmean was calculated for the first and last parts of the curve.
  For the SFI, the part of the curve before the peak force was excluded from the calculation. Within the remaining curve, the area under the force-time curve and a hypothetical area under the force-time curve were calculated. The hypothetical area under the force-time curve mimics a situation in which strength would have been sustained at the maximum level during the trial and no
Dynamic motor fatigability | Baseline, immediately after the intervention and after 2 months follow-up
  Assessed with Biometrics E-LINK H-500 Hand Kit (dynamometer).
  Dynamic motor fatigability will be measured while the child had to squeeze repeatedly as hard and fast as possible during a 30-second period. The measurement will be successful if the child repeatedly squeezed over the entire 30 seconds regardless of the frequency (Brauers 2022). Three trials of this measurement will be performed.
  Dynamic motor fatigability was quantified by Fmean and the number of peaks (Npeaks). The 30-second force-time curve was divided into 3 equal parts (10 seconds each), and Fmean and Npeaks were calculated for the first and third parts. A decrease in Fmean and/or a decrease in Npeaks between the first and third parts indicated higher motor fatigability.
Hand Dexetrity | Baseline, immediately after the intervention and after 2 months follow-up
  Box and Block Test (BBT) will be used for measuring hand dexterity by using two compartment box containing 150 blocks. The test includes grasping, moving, and releasing wooden blocks from one side to the other. The score was recorded for 1 minute as the number of blocks passed over the wooden partition
Participation measures | Baseline, immediately after the intervention and after 2 months follow-up
  Participation and Environment Measure (Young Children YC-PEM, for 3- to 5-year-old participants; Children PEM-CY, for-5 to 7-years-old participants) will be administered.
  Young Children Participation and Environment Measure (YC-PEM)
  The YC-PEM and PEMCY analyze the child's participation in different contexts, as well as the characteristics and resources of the environment and it´s implication on participation in children with or without disabilities. It´s a questionnaire, that families respond, and which also allows to know their desire of change, and different strategies they use to optimize the child's participation in their activities of daily life.
  Scores are calculated for each setting through: 1) The average of all frequency ratings (range = 0-7) are used to calculate frequency; 2) The average of all involvement ratings (range = 1-5) are used to calculate level of involvement; 3) The number of items scored as "yes, change desired" are added, divided by the total number o
Quality of life measures | Baseline, immediately after the intervention and after 2 months follow-up
  The Pediatric Quality of Life Inventory (PedsQL) cerebral palsy and multidimensional fatigue module, parental version is used.
  It´s a questionnaire that assesses the quality of life of children from 2 to 18 years. It contains a specific module for children with cerebral palsy. Parents can make the report from 2 to 18 years and assessed the perceptions of parents about their children's HRQOL. The scale contains 35 items and covers aspects of daily activities, school, movement and balance, pain, fatigue, eating activities, speech and communication. The scientific literature relating to PedsQL supports the reliability, validity, and sensitivity of the PedsQL in children with cerebral palsy.
Attention measures | Baseline, immediately after the intervention and after 2 months follow-up
  Teddy Bear Cancellation Test will be use to measure selective attention and hemineglect in children with unilateral cerebral palsy. A digital version of Teddy Bear is used to obtain more data of the assessment.
Self-perceived occupational performance | Baseline, immediately after the intervention and after 2 months follow-up
  The Canadian Occupational Performance Measure (COPM) will be used to assess the children's self-perceived occupation performance over different categories, including self-care, leisure and productivity. The parents or caregiver rates performance and satisfaction for each functional goal on a ten point ordinal scale, where 1 = "not able to do it all"/"not satisfied at all" and 10 = "able to do it extremely well"/"extremely satisfied".
Goal attainment | Baseline, immediately after the intervention and after 2 months follow-up
  Goal attainment will be objectified using the Goal Attainment Scale (GAS) for at least two individualized therapy goals. The GAS enables the conversion of goal attainment on a 5-point scale into t-scores. The score for each functional outcome ranges from -3 to 2. The participant's baseline performance is represented by a score of -2. Improvements in functional goal performance correspond to scores ranging from -1 to +2, with score 0 being the expected outcome.
Usability measures | immediately after the intervention
  Subjective Usability Scale (SUS), a Likert-type scale with questions about effectiveness (can users achieve their objectives), efficiency (how much effort is expending in achieving the objectives) and satisfaction while using the WeFun-wearable.
Adherence measures | immediately after the intervention
  In terms of adherence we will register number of weeks participating in the intervention, number and type of activities performed and possible dropouts. For checking acceptability and safety we will register parents´ answers some questions using a Likert-type scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade da Coruña, A Coruña, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Albrecht EC, Khetani MA. Environmental impact on young children's participation in home-based activities. Dev Med Child Neurol. 2017 Apr;59(4):388-394. doi: 10.1111/dmcn.13360. Epub 2016 Dec 17. PMID 27988938
- [Background] Reid LB, Rose SE, Boyd RN. Rehabilitation and neuroplasticity in children with unilateral cerebral palsy. Nat Rev Neurol. 2015 Jul;11(7):390-400. doi: 10.1038/nrneurol.2015.97. Epub 2015 Jun 16. PMID 26077839
- [Background] Gordon AM, Bleyenheuft Y, Steenbergen B. Pathophysiology of impaired hand function in children with unilateral cerebral palsy. Dev Med Child Neurol. 2013 Nov;55 Suppl 4:32-7. doi: 10.1111/dmcn.12304. PMID 24237277
- [Background] Carton de Tournai A, Herman E, Ebner-Karestinos D, Gathy E, Araneda R, Renders A, De Clerck C, Kilcioglu S, Dricot L, Macq B, Vandermeeren Y, Bleyenheuft Y. Hand-Arm Bimanual Intensive Therapy Including Lower Extremities in Infants With Unilateral Cerebral Palsy: A Randomized Clinical Trial. JAMA Netw Open. 2024 Nov 4;7(11):e2445133. doi: 10.1001/jamanetworkopen.2024.45133. PMID 39556397